CLINICAL TRIAL: NCT06072066
Title: The Effects of Oral Supplement Containing L-Histidine and Antioxidants on the Skin Barrier Function and Systemic Inflammation in Rosacea
Brief Title: Effects of Oral Supplement Containing L-Histidine and Antioxidants on the Skin Barrier Function and Systemic Inflammation in Rosacea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Skin Science and Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: i23-04_CL_SkinBarrier_Supp
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Rosacea; Systemic Inflammation
Keywords: Rosacea; L-Histidine; Antioxidants
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin Barrier Oral Supplement (Experimental)
  Interventions: Dietary Supplement: Skin Barrier Oral Supplement

INTERVENTIONS:
Dietary Supplement: Skin Barrier Oral Supplement — Supplment powder

SUMMARY:
The purpose of this study is to evaluate how supplementation will alter the skin and the gut barrier and inflammation in those with rosacea.

DETAILED DESCRIPTION:
Rosacea is a chronic inflammatory condition that widely prevalent in the general population and is associated with both inflammation and dysfunction of the skin barrier. Gut dysfunction has been shown to be present in those with rosacea. This study evaluates how the use of a supplement may improve the gut and skin barrier as well as reduce general inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 30 to 70 years of age
* The presence of mild to moderate rosacea (erythematotelangiectatic or papulopustular)
* High sensitivity C-reactive protein (hs-CRP) that is greater than or equal to 1.0 mg/L

Exclusion Criteria:

* The presence of severe rosacea as noted by the investigator global assessment.
* Those who are unwilling to discontinue oral supplementation, or supplement ingredients found in the study's oral product 1 month prior to enrollment.
* Discontinuation of oral L-glutamine or L-glutamine containing supplement 1 month prior to enrollment
* Those who are unwilling to discontinue topical benzoyl peroxide or retinoids for 2 weeks prior to enrollment.
* Those who are unwilling to keep their facial regimen the same throughout the study.
* Individuals who have been on an oral antibiotic within the previous one month.
* Individuals who are pregnant or breastfeeding.
* Individuals who have changed any of their hormonal based contraception or therapies within 3 months prior to joining the study.
* Individuals on oral contraceptive pills or progesterone or estrogen containing therapies.
* Use of isotretinoin within the three months prior to enrollment.
* Individuals on finasteride or dutasteride
* Current tobacco smoker, smoker within the past year, or greater than 5 pack-year tobacco smoking history.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Transepidermal water loss (TEWL) | 8 weeks
  Change in the facial transepidermal water loss (TEWL) using the Vapometer.
Blood hs-CRP level | 8 weeks
  Change in blood hs-CRP level through blood spot testing

SECONDARY OUTCOMES:
Intestinal permeability | 4 weeks
  Change in intestinal permeability through a urine based test by Genova Diagnostics
Intestinal permeability | 8 weeks
  Change in intestinal permeability through a urine based test by Genova Diagnostics
Fecal levels of calprotectin | 4 weeks
  Change in fecal levels of calprotectin through a stool sample
Fecal levels of calprotectin | 8 weeks
  Change in fecal levels of calprotectin through a stool sample
Transepidermal water loss (TEWL) | 4 weeks
  Change in the facial transepidermal water loss (TEWL) using the Vapometer.
Blood hs-CRP level | 4 weeks
  Change in blood hs-CRP level through blood spot testing
Mood Questionnaire | 4 weeks
  A survey to assess changes in mood
Mood Questionnaire | 8 Weeks
  A survey to assess changes in mood
Digestive Questionnaire | 4 weeks
  A survey to assess digestive health
Digestive Questionnaire | 8 weeks
  A survey to assess digestive health

OTHER OUTCOMES:
Inflammatory lesions on the face | 4 weeks
  Change in number of inflammatory lesions on the face
Inflammatory lesions on the face | 8 weeks
  Change in number of inflammatory lesions on the face
Facial erythema | 4 weeks
  Change in appearance of facial erythema measured by photographic analysis (BTBP 3D Camera System)
Facial erythema | 8 weeks
  Change in appearance of facial erythema measured by photographic analysis (BTBP 3D Camera System)

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No